CLINICAL TRIAL: NCT02448485
Title: High-Sensitivity Troponin T Plasma Levels in Patients With Aortic Stenosis
Brief Title: High-Sensitivity Troponin T Plasma Levels in Patients With Aortic Stenosis (Tyrolean Aortic Stenosis Study-2)
Acronym: TASS-2
Status: Recruiting | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Wolfgang Dichtl, MD PhD, Priv.-Doz. DDr., Medical University Innsbruck
Other Study IDs: TASS-2
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Aortic Stenosis; Heart Failure; Syncope; Angina Pectoris
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Failure; Syncope; Angina Pectoris | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Aortic Valve Intervention: Consecutive symptomatic patients who underwent aortic valve intervention (SAVR or TAVI) for the treatment of severe AS since 2010
  Interventions: Procedure: Aortic Valve Intervention (surgical or transcatheter)
- Conservative Treatment: Asymptomatic patients with aortic stenosis followed conservatively at our department

INTERVENTIONS:
Procedure: Aortic Valve Intervention (surgical or transcatheter) — Surgical or interventional aortic valve implantation
  Groups: Aortic Valve Intervention

SUMMARY:
TASS-2 (Tyrolean Aortic Stenosis Study-2) aims to characterize the clinical value of minimally elevated troponin T plasma levels both in patients with asymptomatic and symtomatic aortic stenosis.

DETAILED DESCRIPTION:
Development of symptoms such as heart failure, syncope or angina pectoris is the well-established indication for valve operation in patients with severe aortic stenosis. However, many patients tend to misinterpretate or even ignore symptom onset, and irreversible myocardial dysfunction may occur. Measurement of aortic valve area by transthoracic echocardiography using the continuity equation is prone to methological mistakes, whereas transvalvular gradients are usually easy to quantify but may underestimate hemodynamic effects in the presence of low flow (stroke volume index below 35 ml/m2). All these shortcomings in clinical routine may be overcome by objectively and easily assessable parameters indicating advanced aortic stenosis. Severe aortic valve calcification is such a risk factor for worse prognosis. However, assessment of valve calcification by echocardiography is a subjective measurement and highly operator-dependent. Quantification of valve calcification by multi detector computed tomography is limited by exposure to radiation, availibilty and cost.

A laboratory parameter already used in clinical routine would fullfill the requirements for such a risk stratification much better. Natriuretic peptides may be of interest in this context, but their plasma levels are strongly influenced by age, sex, concomitant arterial hypertension and/or renal dysfunction and volume status. Recently, high-sensitivity troponin plasma levels have been suggested to indicate ongoing myocardial fibrosis in aortic stenosis. A small study with 60 patients suggested that hs-TnT predicte the operative outcome of AS. We therefore set out to characterize the clinical value of minimally elevated troponin T plasma levels both in patients with asymptomatic and symtomatic aortic stenosis.

ELIGIBILITY:
Inclusion Criteria:

* aortic stenosis detected by echocardiography / invasively

Exclusion Criteria:

* acute coronary syndrome
* endocarditis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: One patient cohort consists of patients with severe symptomatic aortic stenosis admitted for planned valve operation since 2010, when involved institutions started to routinely analyse hsTnT plasma levels.
  The other patient cohort consists of asymptomatic patients with aortic stenosis diagnosed treated conservatively.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Mortality (overall, cardiovascular) | up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Dichtl, MD, PhD, Principal Investigator — Medical University Innsbruck
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria